CLINICAL TRIAL: NCT06744491
Title: Anabolic Sensitivity Across the Lifespan
Brief Title: Oral 'Breath Test' to Measure Anabolic Sensitivity to a Protein Meal Across the Age and Physical Activity Spectrum
Acronym: NFRF
Status: Not yet recruiting | Type: Observational
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Daniel Moore, Professor, Muscle Physiology, University of Toronto
Other Study IDs: 00044004
Record Dates: First submitted 2024-12-16; First posted 2024-12-20 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-11

CONDITIONS: Inactivity, Physical; Aging; Healthy Aging; Growth & Development; Sex Differences; Anabolic Sensitivity; Protein Metabolism; Physical Activity
Keywords: anabolic sensitivity; aging; growth and development; physical activity; skeletal muscle; stable isotopes
MeSH Terms: conditions — Sedentary Behavior; Motor Activity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Urine and saliva samples will be retained, though not for the purpose of DNA extraction.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Children: Children as defined by maturity offset via age from peak height velocity (aPHV < -1.0 years).
- Adolescent: Adolescents as defined by maturity offset via age from peak height velocity (aPHV -0.5 to +1.5 years)
- Young Adults: Young adults as defined by chronological age between ages 18 - 35 years
- Older Adults: Older adults as defined by chronological age between ages 60 - 80 years

SUMMARY:
The purpose of this study is to determine how anabolic sensitivity, in response to the ingestion of a liquid protein meal, differs across the lifespan, between biological sexes, and with varying physical activity levels.

DETAILED DESCRIPTION:
Skeletal muscle is a dynamic tissue that responds to anabolic (i.e., growth) stimuli such as protein ingestion and exercise. Differences in age and physical activity levels will influence an individual's ability to respond to these anabolic stimuli; this concept is known as anabolic sensitivity. For instance, older and less physically active individuals will display lower anabolic sensitivity (i.e., anabolic resistance) to a bout of exercise or the consumption of protein in comparison to younger, more physically active individuals. Seeing that individuals with anabolic resistance are at a greater risk for losing muscle mass over time, it is important to understand the anabolic sensitivity/resistance of an individual to assess for the efficiency of growth across the health and lifespan, in addition to a potential screen for metabolic alterations that could manifest into changes in lean body and muscle mass.

Traditional methods to assess for skeletal muscle anabolism and protein metabolism requires in-person and invasive research methods (i.e., stable isotope infusions and muscle biopsies) in controlled laboratory or clinical settings. However, there are many risks associated with these invasive procedures and they are not always feasible in all populations (e.g., children, clinical populations, etc..). Our lab has recently developed a non-invasive 13C breath test which employs an oral stable isotope tracer. Our breath test allows us to assess for anabolic sensitivity in response to protein ingestion, by determining how much of the ingested protein was used to build (synthesize) new proteins in our body (i.e., anabolism) or used as a source of energy (through a process called oxidation). As such, the purpose of the present study is to determine how anabolic sensitivity, in response to the ingestion of a liquid protein meal, differs across the lifespan and with varying physical activity levels.

ELIGIBILITY:
Inclusion Criteria:

* Healthy will be defined as screened by the PAR-Q+ (The Physical Activity Readiness Questionnaire for everyone)
* Chronological age for Healthy Young (age: 18-35 years) or Older (age: 60-80 years) adults
* Chronological age between 8 to 16 years, with maturity offset < -1 year from age of Peak Height Velocity (aPHV) for children and between -0.5 to +1.5 years from aPHV in adolescent participants
* BMI between normal to overweight (18.5 - 29.9 kg/m2)

Exclusion Criteria:

* Regular use of nonsteroidal anti-inflammatory dugs (with the exception of daily low-dose aspirin)
* use of anticoagulants
* use of a walker, cane, or assistive walking device
* infectious or gastrointestinal disease
* inability to comply with study protocol (e.g., unable to track diet)
* regular tobacco use
* self-reported illicit drug use (e.g., growth hormone, testosterone, etc.)
* diagnosed chronic illness (e.g., type 2 diabetes, heart disease, thyroid disease)
* pregnant
* hormonal replacement therapy

Ages: 8 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Convenience sample of individuals who qualify for the corresponding cohorts based on inclusion/exclusion criteria stated.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-12-20 (Estimated); Primary Completion 2025-05-30 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Amino acid oxidation and net protein balance | 6 Hours
  Amino acid oxidation and net protein balance assessed by oral 1-13C Leucine tracer. Net protein balance is derived from the difference between amino acid intake (known) and total amino acid oxidation over the 6h post-prandial measurement period.

CONTACTS AND LOCATIONS:
Locations (1):
- Goldring Center for High Performance Sport, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided